CLINICAL TRIAL: NCT05117333
Title: Reminders, Cost Sharing, and Healthcare Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Lauri Sääksvuori, Associate professor, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: THL/3181/6.02.01/2021
Record Dates: First submitted 2021-10-05; First posted 2021-11-11 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Health Care Utilization; Health Care Seeking Behavior; Health Behavior
Keywords: Cost-sharing, primary care, health care utilization
MeSH Terms: conditions — Patient Acceptance of Health Care; Health Behavior

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with three active treatment arms and a control group (not assigned to any treatment, information and services as usual).
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a randomized experiment in which individuals receive different types of reminders. All outcome variables are based on administrative (secondary) data. Individuals receiving letters and care providers are not aware of the experiment. Investigators will not have any contact with the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Basic letter (Active Comparator): This reminder states that if healthcare is not consumed at the right time, health may deteriorate and diagnoses and treatment may be delayed.
  Interventions: Other: Reminder (information letter)
- Co-pay (Active Comparator): This reminder states that if healthcare is not consumed at the right time, health may deteriorate and diagnoses and treatment may be delayed AND informs recipients about a new law that abolished all co-payments for all primary care nurse visits in Finland.
  Interventions: Other: Reminder (information letter)
- GP-Co-pay (Active Comparator): This reminder states that if healthcare is not consumed at the right time, health may deteriorate and diagnoses and treatment may be delayed AND informs recipients about a new law that abolished all co-payments for all primary care nurse visits in Finland, AND informs recipients that the new law did not abolish co-payments related to general practitioner visits.
  Interventions: Other: Reminder (information letter)
- Control treatment (No Intervention): There is no intervention in the control treatment. The entire population aged 55 and above in the treatment regions will serve as a control group.

INTERVENTIONS:
Other: Reminder (information letter) — Reminders
  Arms: Basic letter; Co-pay; GP-Co-pay

SUMMARY:
The investigators conduct a large-scale randomized controlled trial in Finland by sending three types of information letters to households to examine whether the reminder letters affect healthcare use. All letters remind of the importance of seeking care to treat potential health problems.

This study has two primary objectives are: to evaluate the effects of an information nudge reminding on the importance of diagnosing and treating health problems and to evaluate the effects of additionally providing information on the fact that primary care nurse visits have become exempt from copayments. Main outcomes include the number of primary care nurse visits and general practitioner (GP) visits in a six-month follow-up.

DETAILED DESCRIPTION:
This study has two main objectives: (i) to evaluate the effect of an information nudge reminding on the importance of diagnosing and treating health problems and (ii) to evaluate the effect of providing information on the fact that primary care nurse visits have become exempt from co-payments.

ELIGIBILITY:
Inclusion Criteria:

* Residency in one of the 25 target municipalities as of September 15, 2021.
* Born in 1966 or earlier (aged 55 or more at the end of 2021).
* Living in a household with a maximum of three individuals aged 55 or above.

Exclusion Criteria:

* Individuals living in households (postal address) with more than three individuals aged 55 and above.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47398 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of nurse visits (as recorded in the Finnish National Register of Primary Health Care Visits) | Six months starting from the date the letters are sent
Number of doctor visits (as recorded in the Finnish National Register of Primary Health Care Visits) | Six months starting from the date the letters are sent

SECONDARY OUTCOMES:
Number of referrals to specialized care (as recorded in the Finnish National Register of Primary Health Care Visits) | Six months starting from the date the letters are sent
Number of drug prescriptions for newly initiated therapies (as recorded in the Finnish national register for prescribed medicines) | Six months starting from the date the letters are sent

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Sääksvuori, PhD, Principal Investigator — Finnish Institute for Health and Welfare and University of Turku
Locations (1):
- Finnish Institute for Health and Welfare, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
This paper uses administrative health records maintained by the Finnish Institute for Health and Welfare. Access to health records is regulated in Finland under the Act on the Secondary Use of Health and Social Data (552/2019). De-identified individual participant data will be shared subject to approval by the competent data protection authority. All statistical code used to organize and analyze the data will be shared.